CLINICAL TRIAL: NCT06626672
Title: Digital Lifestyle Intervention to Promote Physical Activity, Nutrition, and Health Literacy in Children With Congenital Heart Disease and Their Guardians
Brief Title: Digital Health Promotion for Children With Congenital Heart Disease and Their Guardians
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Deutsches Herzzentrum Muenchen (Other)
Collaborators: Technical University of Munich (Other); Stiftung KinderHerz Deutschland gGmbH (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2024-337-S-SB
Record Dates: First submitted 2024-10-02; First posted 2024-10-04 (Actual); Last update posted 2025-01-29 (Actual); Status verified 2025-01

CONDITIONS: Congenital Heart Disease; Pediatric ALL
Keywords: Congenital Heart Disease; Congenital Heart Defect; Child; Physical Activity; Exercise; MVPA; Digital Health; Telemedicine; Health literacy; Quality Of Life
MeSH Terms: conditions — Heart Defects, Congenital; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Motor Activity

STUDY DESIGN:
Intervention Model Description: The study uses a delayed start design with two arms. In Arm 1, participants receive the intervention immediately for 12 weeks. In Arm 2, participants initially do not receive the intervention but will start the same intervention after a 12-week delay to ensure fairness.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Digital Health Intervention (Experimental): Children and their guardians are given access to a 12-week digital platform with content to improve their lifestyle.
  Physical activity is monitored with a Garmin Vivofit Jr. 2.
  Interventions: Behavioral: Digital Health Intervention
- Control (No Intervention): During 12-week control period participants receive no access the digital platform. Physical activity is monitored with a Garmin Vivofit Jr. 2.

INTERVENTIONS:
Behavioral: Digital Health Intervention — Access to a digital platform including weekly workout videos, live workouts, recipes, study summaries, and a consultation hour.
  Arms: Digital Health Intervention

SUMMARY:
Congenital heart disease (CHD) affects approximately 1% of live births, and children with CHD often fail to meet WHO physical activity guidelines. Digital interventions to promote physical activity in CHD patients are limited. This study will develop and test a 12-week digital lifestyle intervention for children (ages 8-13) and their guardians, using a Garmin Vivofit Jr. 2 wearable to continuously monitor physical activity (PA). We will assess its impact on children's moderate to vigorous intensity physical activity (MVPA), daily activity (steps per day), quality of life, nutrition, and health literacy, as well as the quality of life and health literacy of their parents.

ELIGIBILITY:
Inclusion Criteria:

* Ages 8-14 years
* Presence of a congenital heart defect (must be moderate or complex according to ACC criteria)
* NYHA Class I or II
* Presence of written informed consent

Exclusion Criteria:

* Cognitive impairments that inhibit patients from understanding the tasks
* No sports clearance by paediatric cardiologists

Ages: 8 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2024-10-01 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Physical activity | 12 weeks
  Physical activity is objectively assessed with the wrist worn wearable "Garmin vivofit jr. 2". Daily physical activity is measured on the basis of active minutes in moderate-to-vigorous intensity.

SECONDARY OUTCOMES:
Daily step count | 12 weeks
  Children's daily step count is objectively assessed using the wrist-worn wearable device, Garmin Vivofit Jr. 2.
Health-related quality of life | Baseline, after 6 weeks, after 12 weeks
  Children's health-related quality of life is self-assessed via the KINDL® questionnaire. The KINDL® is a generic instrument for assessing health-related quality of life in children and adolescents. The KINDL® is a short, methodologically tested and flexible measurement instrument consisting of 24 questions on the six areas of body/physis, feelings/psychology, self-assessment, family, friends and school.
Physical Activity Health Literacy | Baseline, after 6 weeks, after 12 weeks
  Physical Activity Health Literacy Scale for Children (PAHL-C) evaluates children's self-reported knowledge and understanding of physical activity and its benefits through an 8-question scale.
Nutritional Health Literacy | Baseline, after 6 weeks, after 12 weeks
  The Nutrition Health Literacy Scale for Children (NHL-C) measures children's self-reported knowledge and understanding of nutrition and healthy eating using an 8-question scale.
Health-Related Quality of Life: Parent Version (Proxy-Report) | Baseline, after 6 weeks, after 12 weeks
  The KINDL® proxy-report assesses the child's health-related quality of life from the parent's perspective, using the KINDL® questionnaire designed for parents to provide insights on the child's health-related quality of life.
Health Literacy for Children | Baseline, after 6 weeks, after 12 weeks
  Health Literacy Survey Questionnaire for Children (HLS-Child-Q15) assesses children's ability to seek, evaluate, and use health information, including disease prevention and health promotion.
Health Literacy for Adults | Baseline, after 6 weeks, after 12 weeks
  Health Literacy Questionnaire (HLS EU-Q16) measures general health literacy in adults, covering access, understanding, and application of health information across various health domains.

CONTACTS AND LOCATIONS:
Overall Officials: Jan Müller, Prof. Dr., Principal Investigator — Technical University of Munich, Chair of preventive perdiatrics
Locations (1):
- Department of Paediatric Cardiology and Congenital Heart Defects, German Heart Center of the State Bavaria (Munich), Technical University of Munich (TUM), München, Germany

IPD SHARING:
Plan to Share IPD: No